CLINICAL TRIAL: NCT00133393
Title: Dose Finding Study of Pentoxifylline in Children With Cerebral Malaria
Brief Title: Pentoxifylline in Children With Malaria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-021
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-10

CONDITIONS: Plasmodium Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline

SUMMARY:
The primary objectives of this study is to identify a safe, tolerable dose of pentoxifylline in children with cerebral malaria and to establish an acceptable pentoxifylline dosage regimen for use in multi center Phase II and Phase III studies.

DETAILED DESCRIPTION:
This is an open, prospective, dose-escalating study, designed to elucidate the pharmacokinetics, pharmacodynamics, safety, and tolerability of pentoxifylline in children of the ages greater than/equal to 9 months and less than/equal to 96 months with cerebral malaria. The study is designed to evaluate pentoxifylline as adjunct therapy in severe pediatric malaria by evaluating its toxicity and associated adverse events, and by establishing both an acceptable dose and the associated pharmacokinetic profile. The pharmacodynamic effects of four different dose levels (10, 20, 30, and 40 mg/kg/24 hours) will be accessed on the following biological, immunological, and parasitological parameters: cerebral blood flow velocity, tumor necrosis factor concentration, rosetting, coma resolution time, parasite clearance time, and fever clearance time. Due to the variability observed in the biological, immunological, and parasitological parameters under scrutiny, a control group of ten patients will be intercalated in the study (4 patients prior to enrollment of the first pentoxifylline recipient, 2 patients in-between each of the 3 dose escalations). As there is no information about the relationship of treatment duration to biological, immunological, and parasitological effects, treatment will continue for 72 hours, by which time peripheral parasitemia will have cleared in the majority of patients. The selection of the pentoxifylline dosage regimen for the larger, multi center Phase II and Phase III studies will be made on the basis of the maximum tolerated dose (based on clinical and laboratory observations) which minimizes the dose-related side-effects and adverse events (based on pharmacokinetics) while permitting maximum biological, immunological, and/or parasitological effects (pharmacodynamics).

ELIGIBILITY:
Inclusion Criteria:

Children meeting all of the following criteria are eligible for inclusion in the study.

Age greater than or equal to 9 months and less than or equal to 96 months. Informed consent granted by parents/guardians (Appendix I).

Has cerebral malaria defined as all of the following:

peripheral parasitemia with asexual forms of P. falciparum; inability to localize a painful stimulus 30 minutes after correcting hypoglycemia (blood glucose less than 2.2 mmol/l) in patients who present with hypoglycemia 30 minutes after cessation of convulsive activity in patients who are convulsing on admission; no neck stiffness; no clinical evidence of pneumonia (no rales, no decreased breath sounds, no bronchial breathing).

Exclusion Criteria:

Children with the following will not be enrolled in the study:

Hypotension: mean blood pressure less than 60 mmHg (mean blood pressure = diastolic blood pressure (mmHg) + 1/3 (systolic blood pressure

* diastolic blood pressure)). Thrombocytopenia: platelet count less than 50 x 10(to the ninth power)/l. Spontaneous bleeding noted in mouth, throat, nares, rectum, or a venipuncture site following adequate pressure.

Hematocrit < 20% OR hematocrit between 20-25% with parasitemia greater than 10%.

Ages: 9 Months to 96 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2002-01; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI Centre for Geographic Medicine Research, Kilifi, Kenya